CLINICAL TRIAL: NCT04675190
Title: History of Abdominal Surgery Can be a Risk Factor of Gall Stone Disease? A Case Control Study
Brief Title: Major Surgery as a Risk of Gall Stone Disease?
Status: Completed | Type: Observational
Sponsor: Nepal Medical College and Teaching Hospital (Other)
Collaborators: Lumbini Medical College (Other); Chitwan Medical College (Other)
Responsible Party: Principal Investigator, Nabin Pokharel, Associate Professor, Nepal Medical College and Teaching Hospital
Other Study IDs: 024-077/078
Record Dates: First submitted 2020-12-04; First posted 2020-12-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Gall Stones (& [Calculus - Gall Bladder]); Surgery
Keywords: Abdominal Surgery; Gall Stones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Case: Cases will be patients in the department of surgery above 18 years with ultrasound findings of gall stone disease.
  Interventions: Procedure: Major abdominal Surgery
- Control: Controls will be patients in the department of surgery above 18 years with ultrasound findings showing evidence of no gallstones
  Interventions: Procedure: Major abdominal Surgery

INTERVENTIONS:
Procedure: Major abdominal Surgery — Any surgery performed under general or regional anesthesia and procedures involving abdominal cavity is considered major abdominal surgery and those who have undergone any major abdominal surgery before 6 months from the date of ultrasound findings confirming the presence or absence of gall stone will be considered exposed.

SUMMARY:
Gall stone disease is one of the most common diseases occurring in the world as well as in our country, Nepal. This disease is problematic to a lot of patients and poses a huge economic burden to the country. Gall stone disease is usually diagnosed by abdominal ultrasonography as echogenic foci that cast an acoustic shadow. The risk factors for the development of gall stones are multiple; age, sex, genetic susceptibility, pregnancy, dyslipidemia, obesity, rapid weight loss, prolonged fasting and parenteral nutrition, spinal cord injury, cirrhosis, hyperbilirubinemia, and Crohn's disease. In cases of prolonged fasting, total parenteral nutrition, and spinal cord injury; biliary stasis due to lack of enteral stimulation is thought to contribute for the development of gall stones.8 Biliary stasis leads to the formation of sludge which consists of mucus, calcium bilirubinate, and cholesterol crystals. It has been established that several drugs viz.fibrates, ceftriaxone, somatostatin analogues and oral contraceptive pill can promote gall stone formation.

The elective surgeries are performed after preoperative fasting >6 hrs. as recommended by different society of anesthesiology. Moreover, fasting continues throughout surgery and few post-operative hours which usually lasts more than 12 hours. Also group of people after major abdominal surgeries frequently develop post-operative hyperbilirubinemia.

All these factors after any major surgeries may pose a risk for the development of Gall stones.

The major goal of this study is to look if the history of major surgery in the past is one of the etiological factors for the development of gall stone disease. It is a case-control study carried out in the Department of Surgery. It will also help us analyze other multiple epidemiological factors like age, sex, BMI, drugs, lipid profile, family history lifestyle, and dietary factors associated with the disease. The epidemiological data from this study can also help us analyze other confounding and determining factors.

DETAILED DESCRIPTION:
The risk factors for the development of gall stones are multiple which a reason for its high prevalence. Past history of major surgeries does carry some of the biological causations of the gall stones like prolonged fasting during the perioperative period and post-operative hyperbilirubinemia, effects of stress in the gall bladder, and bile flow. However, there have not been recent studies to redefine the etiology of gall stone and history of major surgery. Meanwhile, some of the studies are found be of a great value for the background of this study.

A study published by J M Little and J Ivramovic in 1991 showed that the major abdominal surgery had a statistically significant difference in a cumulative prevalence of the gall stone compared to those who did not undergo any surgery. However, the exact mechanism behind the formation of the stone was not revealed but the sludge formation during fasting was assumed to be the common pathways. L Bolondi, S Gaiani have ultrasonographically assessed the prevalence of sludge in a group of 48 fasting patients after gastrointestinal tract surgery with a period of fasting lasting for 7 to 10 days. It showed the presence of gall stones with different ultrasonographic patterns in three sludge positive patients after the end of six months. They concluded in the early postoperative period there is a high risk for sludge development and that in some cases sludge may subsequently evolve into gall stones.

Another cross-sectional study by A F Attili,E Scafato showed that Prevalence of gallstone was higher among subjects who had an overnight fasting period of over 12 hours than subjects with that of less than 12 hours. H M Bloch et al studied the effects of fasting and composition of gall bladder, where the mean cholesterol saturation index was significantly greater after a 15 hour fast (1.35+0.08) than after a 10 hour fast (105+0.10). The cholesterol saturation index is the ratio of the cholesterol of the sample to the maximum soluble cholesterol of that sample. In the study, it was determined by using the criteria of Hegardt and Dam. The saturation index of greater than 1 represents the cholesterol is supersaturated and forms gall stones. Henceforth, the findings suggested that fasting for between 10 to 20 hours increases the risk for gallstones formation. Another study by Lee et al where they followed the 94 patients with biliary sludge for the mean of 37.8 months. It was found that 8.3% developed asymptomatic gall stones and 6.3% underwent cholecystectomy.

Another prospective study by Christine Evans et al followed 180 patients following major operations found an incidence of 3.7% severe jaundice and 16.5% mild jaundice (serum bilirubin 1.5-4 mg/dl) and a study by Stefan Stenderet al followed 61,212 patients for 34 years, which showed that the risk for gall stone disease is significantly higher in population with bilirubin level in 10th decile (geometric mean 1.34 gm/dl). Though the previous studies have examined the relationship between fasting and the formation of gallstones, none of them examined the direct relationship between any major surgeries and the incidence of gallstones. They also did not study the other factors like the effects of stress, drugs during surgeries and anesthesia on the gall bladder, and the bile flow. However, they have given enough background to establish a hypothesis that any major surgery can be a significant risk factor for the development of gallstones. However, there is no widely accepted consensus on the grading of surgery so by major surgery we mean all surgeries done under general or regional anesthesia and involves procedures in abdominal cavity.

With our observation of the evidence, it indicates that any major surgery may itself is an important determinant of the gallstone formation soon after the surgery and so a study can address this gap of the knowledge. A case-control study can help us assess the past history of major surgery as a significant risk factor for gallstone disease. Any significant findings will warrant other higher studies like cohort study for a detailed assessment of the cause. It has been evident that prolonged fasting or fasting over 10-12 hours imposes a risk factor for gallstone disease. It has also been established that major gastrointestinal surgery, hyperbilirubinemia is also a risk factor for gallstone disease. However, there is a clear gap of knowledge whether any major surgery with similar biological causation imposes a risk factor for gallstone disease or not. The rationale of the study is to look over this lack of knowledge.

The gall stone disease is itself a major economic burden to a lot of patients and the development of symptomatic gallstone in patients who have undergone major surgery in the past few years would be distressing to the patients and relatives. Even if few people after major surgery develop gall stones in future, and those at such risks could be identified, then we could institute surveillance ultrasonography or medical prophylactic measures like ursodeoxycholic acid.

ELIGIBILITY:
Inclusion Criteria:

* Must be above 18 years of age.

Exclusion Criteria:

* Liver Cirrhosis
* Hepatobiliary and pancreatic malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients above 18 years in the department of surgery in Nepal medical college and teaching hospital, Lumbini Medical College and teaching hospital and Chitwan medical college and teaching hospital
Sampling Method: Probability Sample
Enrollment: 755 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Odds ratio | 2 months
  Ratio of the odds for gall stone disease among patient with past history of major abdominal surgery to patient without history of major abdominal surgery and it its significance.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Dr Katwal, MS, Principal Investigator — Chitwan Medical college and teaching hospital, Nepal; Neeraj Dr. Thapa, MS, Principal Investigator — Lumbini Medical college and teaching hospital, Nepal; Sunil Prof. Dr. Shrestha, MS, Study Chair — Nepal medical college and teaching hospital, Nepal; Harish C Prof. Dr. Neupane, MS, Study Chair — Chitwan Medical college and teaching hospital, Nepal; Kishor K Prof. Dr. Tamrakar, MS, Study Chair — Chitwan Medical colllege and teaching hospital, Nepal; Nabin Dr. Pokharel, MCh, Principal Investigator — Nepal medical college and teaching hospital, Nepal; Biplov Dr. Adhikari, MBBS, Study Chair — Nepal medical college and teaching hospital, Nepal
Locations (3):
- Nepal (3):
  - Chitwan Medical college and teaching hospital, Bharatpur, Bagmati
  - Nepal Medical College and teaching hospital, Kathmandu, Bagmati
  - Lumbini Medical College and teaching hospital, Pālpāthok, Lumbini

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Little JM, Avramovic J. Gallstone formation after major abdominal surgery. Lancet. 1991 May 11;337(8750):1135-7. doi: 10.1016/0140-6736(91)92796-5. PMID 1674022
- [Background] Bolondi L, Gaiani S, Testa S, Labo G. Gall bladder sludge formation during prolonged fasting after gastrointestinal tract surgery. Gut. 1985 Jul;26(7):734-8. doi: 10.1136/gut.26.7.734. PMID 3894170
- [Background] Attili AF, Scafato E, Marchioli R, Marfisi RM, Festi D. Diet and gallstones in Italy: the cross-sectional MICOL results. Hepatology. 1998 Jun;27(6):1492-8. doi: 10.1002/hep.510270605. PMID 9620318
- [Background] Bloch HM, Thornton JR, Heaton KW. Effects of fasting on the composition of gallbladder bile. Gut. 1980 Dec;21(12):1087-9. doi: 10.1136/gut.21.12.1087. PMID 7461468
- [Background] Hegardt FG, Dam H. The solubility of cholesterol in aqueous solutions of bile salts and lecithin. Z Ernahrungswiss. 1971 Apr;10(3):223-33. doi: 10.1007/BF02020933. No abstract available. PMID 5104113
- [Background] Lee SP, Maher K, Nicholls JF. Origin and fate of biliary sludge. Gastroenterology. 1988 Jan;94(1):170-6. doi: 10.1016/0016-5085(88)90626-9. PMID 3275565